CLINICAL TRIAL: NCT02135458
Title: Clinical and Medico-economic Assessment of Conventional Care Plus the "Autonom@Dom" Telemonitoring System Versus a Conventional Care Package Alone, for People With Heart Failure in Several French Structures.
Brief Title: Evaluation of the AUTONOM@DOM Telemonitoring System for People With Heart Failure
Acronym: AUTONOM@DOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Medico-economic evaluation unit , University Hospital, Grenoble (Unknown)
Responsible Party: Principal Investigator, AdministrateurCIC, Dr Yannick NEUDER, University Hospital, Grenoble, University Hospital, Grenoble
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DCIC 13 61
Record Dates: First submitted 2014-04-09; First posted 2014-05-12 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure
Keywords: Heart failure; Telemonitoring; therapeutic education; care network; hospitalization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemonitoring (Experimental): Home-based patient management using AUTONOM@DOM telemonitoring system to record and transmit heart rate, blood pressure and weight; along side conventional care (patient therapeutic education or personalised care program)
  Interventions: Other: Telemonitoring; Other: Conventional care
- Conventional care (Active Comparator): Conventional care including patient therapeutic education or personalised care program
  Interventions: Other: Conventional care

INTERVENTIONS:
Other: Telemonitoring
  Arms: Telemonitoring
Other: Conventional care
  Other Names: Patient therapeutic education: ETICS HPGM; or; Personalized care program: RESIC 38

SUMMARY:
Heart failure is the principle cause of hospitalisation for people over 65. the assumption is that a system of home based telemonitoring can reduce the rate of unscheduled hospitalisation or rehospitalisation for heart failure (compared to a care package alone), This randomised controlled pilot study should assess the feasibility in terms of patient inclusion and follow-up.

DETAILED DESCRIPTION:
Chronic diseases such as heart failure are a major burden for healthcare systems They are punctuated by exacerbations, often markers of poor prognosis, and are associated with expensive unscheduled hospitalizations. After initial diagnosis, despite the development of both drug and physical therapies, the rate of re-hospitalization for heart failure remains high with 50% or more of patients readmitted within 6 months.

Recommendations for the treatment of heart failure patients are extremely precise and justify close collaboration between local community services and the hospital. However there is often considerable divergence between recommended care and the reality, due in particular to the difficulty in monitoring ambulatory patients. For example, the dose titration of beta-blockers or ACE inhibitors need to be monitored, and dosages of diuretics need to be adapted to avoid side effects which affect the quality of life of patients and limit medication adherence etc. The establishment of 'ambulatory' care networks (including multidisciplinary health professionnals of city and hospital and therapeutic patient education) such as that in Isère County in France has demonstrated its effectiveness.

However, more advanced tools for patient monitoring still need to be assessed, particularly 'home monitoring', because there is not yet consensus as to the role tele-monitoring should play in the context of heart failure, and to date recommendations are vague. Assess the clinical and medico-economic benefit of an innovative patient monitoring strategy 'AUTONOM @ DOM' is needed.

The primary aim of this study is then to assess a system of home based telemonitoring .The main outcome is unscheduled hospitalisation for heart failure. secondary aims were to assess the efficacy of this system, quality of life and medico-economic benefit.

This pilot study is realised in the Isère and Essonne counties of France. Patients diagnosed with heart failure will be randomized to one of the following groups:

* conventional care including at least a patient education program (ETICS program in Essone county and RESIC38 network in Isere county);
* conventional care, plus home telemonitoring including a recording of the heart rate, blood pressure and weight, remotely transmitted to the cardiologist by an approved validated system that includes an alert monitoring feature.

The study will last one year starting in April 2014.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or more
* Covered by French social security system or equivalent
* Written informed consent signed by patient
* Heart failure diagnosed by a cardiologue
* NYHA stage II, III or IV
* Able to be followed-up for 1 year
* Attend general healthcare education sessions

Exclusion Criteria:

* Freedom restricted by judicial order
* Under legal protection
* Require peritoneal dialysis or hemofiltration
* Participation refused by patient, primary care physician or cardiologist
* Present a severe comorbidity with poor short-term prognosis
* Present asymptomatic heart failure NYHA stage I
* Programmed surgical intervention: valve prosthesis or revascularization
* Impossibility to follow a program of patient education
* Residing in medicalized care facility for persons without autonomy
* Residing outside the recruitment zones

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Hospitalization | one year
  Hospitalization at any time during follow-up, emergency, unplanned, inappropriate or early (within one month) rehospitalization or not.
  The type and length of hospital stay will be recorded.

SECONDARY OUTCOMES:
Comparison of quality of life | one year
  loss of autonomy and loss of function, quality of life, depression and anxiety, malnutrition, mortality and clinical stage of the disease
medicoeconomic criteria | one year
  health expenditures and quality of life first. If follow-up turns out feasible, cost-effectiveness and cost-utility ratios
efficacy telemonitoring system criteria | one year
  number and type of telemonitoring alerts and their clinical relevance

CONTACTS AND LOCATIONS:
Overall Officials: Muriel SALVAT, MD, Principal Investigator — University Hospital, Grenoble
Locations (3):
- France (3):
  - Private Geriatric Hospital Magnolias, Ballainvilliers
  - Hospital Group Mutualiste, Grenoble
  - University Hospital of Grenoble, Grenoble

REFERENCES:
- [Background] Maggioni AP, Greene SJ, Fonarow GC, Bohm M, Zannad F, Solomon SD, Lewis EF, Baschiera F, Hua TA, Gimpelewicz CR, Lesogor A, Gheorghiade M; ASTRONAUT Investigators and Coordinators. Effect of aliskiren on post-discharge outcomes among diabetic and non-diabetic patients hospitalized for heart failure: insights from the ASTRONAUT trial. Eur Heart J. 2013 Oct;34(40):3117-27. doi: 10.1093/eurheartj/eht342. Epub 2013 Sep 2. PMID 23999456
- [Background] Gheorghiade M, Bohm M, Greene SJ, Fonarow GC, Lewis EF, Zannad F, Solomon SD, Baschiera F, Botha J, Hua TA, Gimpelewicz CR, Jaumont X, Lesogor A, Maggioni AP; ASTRONAUT Investigators and Coordinators. Effect of aliskiren on postdischarge mortality and heart failure readmissions among patients hospitalized for heart failure: the ASTRONAUT randomized trial. JAMA. 2013 Mar 20;309(11):1125-35. doi: 10.1001/jama.2013.1954. PMID 23478743
- [Background] Logeart D, Isnard R, Resche-Rigon M, Seronde MF, de Groote P, Jondeau G, Galinier M, Mulak G, Donal E, Delahaye F, Juilliere Y, Damy T, Jourdain P, Bauer F, Eicher JC, Neuder Y, Trochu JN; Heart Failure of the French Society of Cardiology. Current aspects of the spectrum of acute heart failure syndromes in a real-life setting: the OFICA study. Eur J Heart Fail. 2013 Apr;15(4):465-76. doi: 10.1093/eurjhf/hfs189. Epub 2012 Nov 27. PMID 23186936
- [Background] Jourdain P, Juilliere Y; Steering and Working Group Committee Members of the French Task Force on Therapeutic Education in Heart Failure. Therapeutic education in patients with chronic heart failure: proposal for a multiprofessional structured programme, by a French Task Force under the auspices of the French Society of Cardiology. Arch Cardiovasc Dis. 2011 Mar;104(3):189-201. doi: 10.1016/j.acvd.2010.12.003. No abstract available. PMID 21634217
- [Background] Roncalli J, Mouquet F, Piot C, Trochu JN, Le Corvoisier P, Neuder Y, Le Tourneau T, Agostini D, Gaxotte V, Sportouch C, Galinier M, Crochet D, Teiger E, Richard MJ, Polge AS, Beregi JP, Manrique A, Carrie D, Susen S, Klein B, Parini A, Lamirault G, Croisille P, Rouard H, Bourin P, Nguyen JM, Delasalle B, Vanzetto G, Van Belle E, Lemarchand P. Intracoronary autologous mononucleated bone marrow cell infusion for acute myocardial infarction: results of the randomized multicenter BONAMI trial. Eur Heart J. 2011 Jul;32(14):1748-57. doi: 10.1093/eurheartj/ehq455. Epub 2010 Dec 2. PMID 21127322
- [Background] Jondeau G, Neuder Y, Eicher JC, Jourdain P, Fauveau E, Galinier M, Jegou A, Bauer F, Trochu JN, Bouzamondo A, Tanguy ML, Lechat P; B-CONVINCED Investigators. B-CONVINCED: Beta-blocker CONtinuation Vs. INterruption in patients with Congestive heart failure hospitalizED for a decompensation episode. Eur Heart J. 2009 Sep;30(18):2186-92. doi: 10.1093/eurheartj/ehp323. Epub 2009 Aug 30. PMID 19717851